CLINICAL TRIAL: NCT07302204
Title: Efficacy of Aerobic Exercise Versus Therapeutic Exercises on Exercise-induced Hypoalgesia in Knee Osteoarthritis. Randomized Clinical Trial
Brief Title: Efficacy of Aerobic Exercise Versus Therapeutic Exercises on Exercise-induced Hypoalgesia in Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Cid André Fidelis de Paula Gomes, Professor Phd, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 93560425.7.0000.5511
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise; Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Group (AEG) (Experimental): Participants allocated to the Aerobic Exercise Group (AEG) will perform supervised cycling on an electromagnetic recumbent stationary bicycle three times per week for ten weeks, with at least 24 hours between sessions. Each session will be structured as five minutes of warm up, a progressively longer work phase, and five minutes of cool down. Exercise intensity will be prescribed and monitored using the 6 to 20 Borg Rating of Perceived Exertion scale, targeting light to moderate exertion during warm up and cool down and moderate to somewhat hard exertion during the work phase. Cadence will be maintained around 60 to 80 revolutions per minute and the resistance level will be adjusted to keep participants within the target exertion zone.
  Interventions: Other: Aerobic Exercise
- Therapeutic Exercise Group (TEG) (Active Comparator): Participants allocated to the Therapeutic Exercise Group will receive an individually supervised, land based therapeutic exercise program focusing on warm up, resisted strengthening, neuromuscular training, mobility and balance. Sessions will be performed three times per week for ten weeks, with at least 24 hours between sessions, and will last approximately 60 minutes. Therapeutic exercises will be completed in up to three sets of 8 to 12 repetitions in weeks 1 to 5 and 8 to 15 repetitions in weeks 6 to 10, each set lasting 30 to 60 seconds, with 90 second rest intervals between sets. Load for machine or free weight exercises will be prescribed at about 40 to 60 percent of the pain limited one repetition maximum, elastic band resistance will be set to allow 12 repetitions with pain ≤ 5 out of 10, and body weight exercises will be held for 30 to 60 seconds. Vital signs and knee pain intensity will be assessed before, during and after each session to guide safety and progression.
  Interventions: Other: Therapeutic Exercise

INTERVENTIONS:
Other: Aerobic Exercise — Supervised cycling on an electromagnetic recumbent stationary bicycle three times per week for ten weeks, with at least 24 hours between sessions.
  Arms: Aerobic Exercise Group (AEG)
Other: Therapeutic Exercise — Individually supervised, land based therapeutic exercise program focusing on warm up, resisted strengthening, neuromuscular training, mobility and balance.
  Arms: Therapeutic Exercise Group (TEG)

SUMMARY:
The study compares two exercise strategies in people with knee osteoarthritis. The first is aerobic exercise on a recumbent cycle ergometer, with effort controlled by the Borg scale. The second is a therapeutic exercise program with resistance, neuromuscular, mobility, and balance components. The primary objective is to determine which approach produces greater exercise induced hypoalgesia, measured by the increase in pressure pain threshold at the knee within the session across four anchor sessions during a ten week program. This is a randomized clinical trial with two parallel arms. Ninety participants, between forty five and seventy five years of age, will be allocated to one of the two groups. Allocation sequence concealment will be ensured using opaque envelopes. The outcome assessor will remain blinded to group allocation. The interventions will take place three times per week for ten weeks. Assessments will be performed at baseline and after ten weeks. Within session measurements will also be taken in weeks one, four, seven, and ten. The primary outcome is the intra session change in pressure pain threshold at the medial compartment of the knee. Secondary outcomes include exercise induced hypoalgesia in the quadriceps and trapezius, chronic adaptation of pressure pain threshold, conditioned pain modulation, pain intensity, pain self efficacy, knee related health status, functional performance, quadriceps strength, global perceived effect, and adherence. The planned sample size is forty five participants per group. The analysis will follow the intention to treat principle. The primary outcome will be compared using linear mixed models with group and time effects. Clinical outcomes at T1 will be adjusted for baseline values. Estimates, confidence intervals, and interpretation in light of minimally important differences will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of symptomatic knee osteoarthritis for at least 3 months.
* Report of knee pain for more than 3 months and average knee pain intensity ≥ 3 on the 0 to 10 Numeric Rating Scale.
* Morning stiffness lasting less than 30 minutes.
* Clinical signs compatible with knee osteoarthritis. crepitus, bony tenderness and absence of palpable warmth at the knee.

Exclusion Criteria:

* Signs and symptoms indicating the hip as the main source of pain.
* Osteoporosis
* Fibromyalgia
* History of tumors or cancer
* Active inflammatory joint diseases, such as rheumatoid arthritis or gout.
* Previous arthroplasty of any lower limb joint.
* Neurological diseases, including Parkinson's disease, stroke, multiple sclerosis, muscular dystrophy, motor neuron disease or Alzheimer's disease.
* Cardiovascular diseases for which exercise is formally contraindicated.
* Infected wounds or osteomyelitis in the knee region.
* Deep vein thrombosis or thrombophlebitis.
* Sensory alterations in the lower limbs.
* Cognitive or cardiopulmonary impairments that limit safe participation in the exercise program.
* Use of walking aids.
* Recent knee trauma.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2029-12-20 (Estimated); Study Completion 2029-12-20 (Estimated)

PRIMARY OUTCOMES:
Exercise-induced hypoalgesia (EIH) | At weeks 1, 4, 7, and 10 of the 10 week intervention (within session, pre and immediately post exercise).
  exercise induced hypoalgesia (EIH) of the medial compartment of the knees, measured by the change in pressure pain threshold (Δ PPT)

SECONDARY OUTCOMES:
Exercise induced hypoalgesia of the quadriceps | Within session, immediately before and immediately after the exercise session at weeks 1, 4, 7, and 10 of the 10 week intervention.
  Within session change in pressure pain threshold at the rectus femoris muscle, calculated as post exercise minus pre exercise values and averaged bilaterally, measured with a digital algometer and expressed in kilograms force per square centimeter.
Exercise induced hypoalgesia of the upper trapezius | Within session, immediately before and immediately after the exercise session at weeks 1, 4, 7, and 10 of the 10 week intervention.
  Within session change in pressure pain threshold at the upper trapezius muscle descending portion, calculated as post exercise minus pre exercise values and averaged bilaterally, measured with a digital algometer and expressed in kilograms force per square centimeter.
Chronic adaptation of pressure pain threshold | Baseline and after 10 weeks of intervention.
  Change in pressure pain threshold at the medial compartment of the knee, rectus femoris and upper trapezius between baseline and post intervention, averaged bilaterally and expressed in kilograms force per square centimeter.
Conditioned pain modulation | Baseline and after 10 weeks of intervention.
  Change in the conditioned pain modulation effect assessed by a standardized conditioned pain modulation test, defined as the change in pressure pain threshold at the volar forearm during and after an ischemic conditioning stimulus on the contralateral arm, with pain intensity standardized around four out of ten on a numeric rating scale.
Pain intensity | Baseline and after 10 weeks of intervention.
  Average knee pain intensity over the past seven days at rest and after movement, measured on an eleven-point numeric rating scale from zero (no pain) to ten (worst imaginable pain). Numeric Rating Scale for Pain Intensity. Range 0 to 10, with 0 indicating no pain and 10 the worst pain imaginable. Higher scores indicate greater pain intensity.
Pain self efficacy | Baseline and after 10 weeks of intervention.
  Pain Self Efficacy Questionnaire. Ten items scored 0 to 6 each, total score 0 to 60. Higher scores indicate better outcome, greater pain related self efficacy.
Knee related health status | Baseline and after 10 weeks of intervention.
  Knee Injury and Osteoarthritis Outcome Score. Subscales are transformed to a 0 to 100 score, where 0 represents the worst knee health status and 100 the best. Higher scores indicate better outcome, better knee related health status.
Patient specific functional status | Baseline and after 10 weeks of intervention.
  Patient Specific Functional Scale. Each selected activity is rated from 0 to 10, where 0 means unable to perform the activity and 10 means able to perform as before the problem. The total score is the mean of the three activities, range 0 to 10. Higher scores indicate better outcome, better patient specific functional status.
Functional performance, thirty second sit to stand test | Baseline and after 10 weeks of intervention.
  Number of full sit to stand repetitions completed from a standard height chair in thirty seconds, higher counts reflecting better lower limb strength, dynamic balance and functional performance.
Quadriceps muscle strength | Baseline and after 10 weeks of intervention.
  Maximal voluntary isometric contraction of the quadriceps measured with a handheld dynamometer in a standardized seated position, normalized to body mass and expressed as a percentage, with higher values indicating greater strength.
Global perceived effect | After 10 weeks of intervention.
  Global Perceived Effect scale. Eleven point scale ranging from minus 5, much worse, to 0, no change, to plus 5, completely recovered. Higher scores indicate better outcome, greater perceived recovery.
Adherence to the intervention | Throughout the 10 week intervention period.
  Proportion of attended exercise sessions relative to the thirty planned sessions, calculated as attendance percentage sessions attended divided by sessions planned multiplied by one hundred.

CONTACTS AND LOCATIONS:
Locations (1):
- Cid André Fidelis de Paula Gomes, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No